CLINICAL TRIAL: NCT00657436
Title: Study of Myeloid-related Protein 8/14 and Additional Biomarkers (Multi Marker Approach) for Early Diagnosis and Risk Stratification in Patients Presenting With Acute Chest Pain at the Emergency Department
Brief Title: Myeloid-Related Protein in Evaluation of Acute Chest Pain in the Emergency Departement
Acronym: MyRiAD
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MyRiAD
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Myocardial Ischemia; Acute Coronary Syndrome; Myocardial Infarction; Coronary Occlusion; Coronary Thrombosis
Keywords: Acute Coronary Syndrome; Myocardial Infarction; Coronary Artery Disease
MeSH Terms: conditions — Myocardial Ischemia; Acute Coronary Syndrome; Myocardial Infarction; Coronary Occlusion; Coronary Thrombosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is the evaluation of multiple biomarkers related to acute coronary syndromes, including myeloid-related protein 8/14 (MRP 8/14), along with established clinical markers, for early diagnosis and risk stratification in patients presenting with acute chest pain at the emergency department.

Study hypothesis: MRP 8/14, alone or together with other established or new biomarkers, increases the earliness, sensitivity, and specificity of diagnosing acute coronary syndromes.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the emergency department of the University Hospital Zurich with measurement of troponin during the routine diagnostic evaluation.

Exclusion Criteria:

* Refusal or inability to give informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients - systematic sampling - presenting with acute chest pain at the emergency room in which determination of cardiac biomarkers is indicated for clinical diagnostics
Sampling Method: Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Diagnosis of acute coronary syndrome | Emergency room and/or hospital stay

SECONDARY OUTCOMES:
Incidence of any acute coronary event | 1 year
Morbidity from coronary artery disease | 1 year
Mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Willibald Maier, MD, Principal Investigator — Cardiology, University Hospital Zurich
Locations (1):
- Cardiology, University Hospital, Zurich, Switzerland

REFERENCES:
- [Background] Altwegg LA, Neidhart M, Hersberger M, Muller S, Eberli FR, Corti R, Roffi M, Sutsch G, Gay S, von Eckardstein A, Wischnewsky MB, Luscher TF, Maier W. Myeloid-related protein 8/14 complex is released by monocytes and granulocytes at the site of coronary occlusion: a novel, early, and sensitive marker of acute coronary syndromes. Eur Heart J. 2007 Apr;28(8):941-8. doi: 10.1093/eurheartj/ehm078. Epub 2007 Mar 26. PMID 17387139